CLINICAL TRIAL: NCT00457561
Title: Recombinant Human Erythropoietin Dose, Serum Adiponectin, and All-Cause Mortality in Patients Beginning Hemodialysis
Status: Completed | Type: Observational
Sponsor: Hamamatsu University (Other)
Other Study IDs: 19710808
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Hemodialysis
Keywords: The relationship between all-cause mortality in patients introduced hemodialysis and recombinant human erythropoietin dose and serum adiponectin level

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Decreased body fat mass, possibly mediated through the effects of elevated serum adiponectin levels, may be associated with requirements for higher recombinant human erythropoietin doses and a subsequent worse prognosis in patients beginning hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who started hemodialysis therapy from August 2000 to May 2001 in 11 dialysis centers in the Shizuoka prefecture area, and who survived for more than 3 months after the start of hemodialysis.

Exclusion Criteria:

* Nothing particular.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Naro Ohashi, MD,PhD, Principal Investigator — First Department of Medicine, Hamamatsu University School of Medicine